CLINICAL TRIAL: NCT03096067
Title: Treatment of Patellar Tendinopathy; Influence of Load Magnitude on Clinical Outcome, Tendon Structure and Function
Brief Title: Patellar Tendinopathy - The Effect of Load Magnitude in Exercise-based Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anne-Sofie Agergaard, PhD Student, MSc. in Physiotherapy, PT, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBH131
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Patellar Tendinopathy; Jumper's Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy slow resistance group (Active Comparator): Heavy slow resistance training. Three times weekly for 12 weeks.
  Interventions: Other: Heavy slow resistance training
- Moderate slow resistance group (Experimental): Moderate slow resistance training. Three times weekly for 12 weeks.
  Interventions: Other: Moderate slow resistance training

INTERVENTIONS:
Other: Heavy slow resistance training — Resistance training for knee extensors. The exercise will be performed at 90% of 1 RM and slowly (6 s/repetition).
  Arms: Heavy slow resistance group
Other: Moderate slow resistance training — Resistance training for knee extensors. The exercise will be performed at 55% of 1 RM and slowly (6 s/repetition).
  Arms: Moderate slow resistance group

SUMMARY:
The purpose of this project is to investigate if the magnitude of a loading based 12 weeks rehabilitation regime for patellar tendinopathy influence the clinical outcome, tendon structure and function.

The investigators hypothesize that a greater magnitude (90% of 1RM) of loading will yield a more positive clinical outcome, tendon structure and function in patients with patellar tendinopathy compared to a lower magnitude of loading (55% of 1 RM) when total exercise volume is equal in both groups.

DETAILED DESCRIPTION:
Randomized controlled intervention study with one year follow-up

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral patellar tendinopathy
* Symptoms > 3 months
* Ultrasonographical tendon swelling
* Ultrasonographical hypo-echoic area with doppler
* BMI 18.5-30

Exclusion Criteria:

* Patellar tendinopathy > 12 month
* Previous knee surgery
* Confounding diagnosis to the knee joint
* Diabetes or arthritis
* Previous corticosteroid injection for patellar tendinopathy
* Smoking
* Being elite volleyball players

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Victorian Institute of Sports Assessment - Patella Questionnaire (VISA-P) at 12 wks | 0-12 wks
  Patient reported outcome regarding symptoms, function and the ability to participate in sports

SECONDARY OUTCOMES:
Victorian Institute of Sports Assessment - Patella Questionnaire (VISA-P) | 0 and 6 wks + 1 yr follow up + Long-term follow-up (2-4 yr)
  Patient reported outcome regarding symptoms, function and the ability to
Pain rating on numeric rating scale (NRS) and activity level of sporting activities (h/wk) | 0,6,12 wks + 1 yr follow up + Long-term follow-up (2-4 yr)
  Questionnaire
Tendon thickness and Doppler activity | 0,6,12 wks + 1 yr follow up + Long-term follow-up (2-4 yr)
  Measured by ultrasound
Single-leg decline squat (SLDS) test | 0,6, 12 wks + 1 yr follow up + Long-term follow-up (2-4 yr)
  A reliable patellar tendon pain provocation test, will be used to assess pain during function
Jump test | 0 and 12 wks
  Squat jump and Counter movement Jump will be used to assess patellar tendinopathy caused functional deficits on the injured site compared with the non-injured site
Mechanical properties | 0 and 12 wks
  Synchronized tendon elongation with the use of ultrasonography along with force measures, will be used during voluntary contractions to determine mechanical properties
Muscle strength | 0 and 12 wks
  Maximal muscle strength of the knee extensors is obtained during a maximal voluntary contractions
Tendon dimensions and structure | 0 and 12 wks
  Measured by MRI
Treatment satisfaction | 12 wks + 1 yr follow-up + Long-term follow-up (2-4 yr)
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Magnusson, Professor, Study Director — Bispebjerg Hospital, University of Copenhagen; Anne-Sofie Agergaard, Phd.Student, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Physical and Occupational Therapy / Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agergaard AS, Svensson RB, Malmgaard-Clausen NM, Couppe C, Hjortshoej MH, Doessing S, Kjaer M, Magnusson SP. Clinical Outcomes, Structure, and Function Improve With Both Heavy and Moderate Loads in the Treatment of Patellar Tendinopathy: A Randomized Clinical Trial. Am J Sports Med. 2021 Mar;49(4):982-993. doi: 10.1177/0363546520988741. Epub 2021 Feb 22. PMID 33616456